CLINICAL TRIAL: NCT01177631
Title: Proteomic Analysis of Human Hepatocellular Carcinoma Associated With Portal Vein Thrombosis
Brief Title: Proteomic Analysis of Human Hepatocellular Carcinoma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Far Eastern Memorial Hospital (Other)
Responsible Party: Principal Investigator, Meng-Tzu Weng, Physician, Far Eastern Memorial Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 97068
Record Dates: First submitted 2009-06-02; First posted 2010-08-09 (Estimated); Last update posted 2016-02-05 (Estimated); Status verified 2016-02

CONDITIONS: Carcinoma, Hepatocellular
Keywords: Carcinoma, hepatocellular; Portal vein; Proteomics
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Surgical Procedures, Operative

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Operation — Operation for clinically evaluated resectable hepatocelluar carcinoma. Compare the different expression of protein between tumor, non-tumor and tumor with vascular invasion part.

SUMMARY:
This is a pilot study to evaluate the difference between the protein expression between hepatocellular carcinoma and tumor with vessel invasion in Asian patients with hepatocellular carcinoma.

ELIGIBILITY:
Inclusion Criteria:

Arm A: Hepatocellular carcinoma with vessel invasion:

* hepatocellular carcionoma, pathologic diagnosed.
* image documented vessel invasion, including portal vein thrombosis
* eligible for surgical intervension.

Arm B: hepatocellular carcinoma without vessel invasion:

* hepatocellular carcinoma, pathologic diagnosed or clinical diagnosed according to EASL criteria.
* no vessel invasion on image.

Arm C: Healthy hepatitis carrier:

* patients age >18 years old with hepatitis B or C
* normal liver function.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2009-02; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
Recurrence | one year
  Evidence of clinically definite vascular invasion of hepatocellular carcinoma. Confirmed by operation. Compare the proteomic expression of tumor, non-tumor ans tumor tissue in vascular part.

CONTACTS AND LOCATIONS:
Locations (1):
- Far Eastern Memorial Hospital, Taipei, Taiwan